CLINICAL TRIAL: NCT05388383
Title: Cost-effectiveness Analysis of Robot-assisted Spinal Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beijing Jishuitan Hospital (Other)
Responsible Party: Principal Investigator, Wei Tian, Director, Head of Spine department, Principal Investigator, Beijing Jishuitan Hospital
Other Study IDs: JST-202101
Record Dates: First submitted 2021-01-14; First posted 2022-05-24 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Lumbar Spine Degeneration; Economic Problems; Surgery
Keywords: robot-assisted; spine surgery; cost-effectiveness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- free-hand: spine surgery without robot
- robot-assisted: Robot-assisted open surgery
  Interventions: Device: Ti-robot
- mi: Robot-assisted minimally invasive surgery
  Interventions: Device: Ti-robot

INTERVENTIONS:
Device: Ti-robot — Tianji ROBOT--Orthopedic surgery robot led by Beijing Jishuitan Hospital
  Groups: mi; robot-assisted

SUMMARY:
With the change of lifestyle and the aging of the population, the prevalence of Lumbar disc herniation (LDH) in my country is increasing year by year, and surgery is one of the main ways to treat LDH. Surgical robots have good application prospects in the surgical treatment of patients with lumbar degenerative diseases. Studies have shown that orthopedic robot-assisted surgery has less soft tissue damage, small surgical incisions, less bleeding, high safety, and quick postoperative recovery; it reduces the risk of spinal cord and blood vessel damage that may be caused during manual operations; does not require repeated fluoroscopy To determine the position of the nail, reduce the intraoperative radiation by more than 70%, and reduce the risk of patient infection.

The current clinical research on robotics technology mainly stays in the aspects of accuracy, effectiveness, and safety. If the technology is promoted in clinical applications, the support of health economics evaluation data is urgently needed. This study hopes to apply robot-assisted technology in LDH surgical treatment through observational research design, evaluate the therapeutic effect and treatment cost of robot-assisted surgery and conventional surgery, focus on health economics evaluation, and provide treatment options for patients and medical care in the health sector. The reasonable allocation of resources and the promotion and application of this technology provide data support.

DETAILED DESCRIPTION:
Beijing Jishuitan Hospital is a pioneer in the research and application of orthopedic robotics in my country. At present, it has completed hundreds of orthopedic surgeries using the "Tianji" robotic system, and has completed a number of randomized controlled clinical trials, proving that robot-assisted surgery is effective in bone degenerative diseases Safety and accuracy in surgical treatment. Based on this platform, this research hopes to apply robot-assisted technology in the treatment of patients with lumbar intervertebral disc herniation, evaluate the therapeutic effect and treatment cost of robot-assisted surgery and conventional surgery, and focus on health economics evaluation, and provide treatment options for patients and health departments The reasonable allocation of medical resources and the promotion and application of this technology provide data support.

ELIGIBILITY:
Inclusion Criteria:

* Diagnose lumbar degenerative diseases and lumbar fractures
* single-level lumbar pedicle screw internal fixation
* Sign informed consent

Exclusion Criteria:

* Multi-level lumbar pedicle screw internal fixation
* QCT diagnoses severe osteoporosis (BMD <60mg/cm3).
* Combined with abnormal coagulation function
* Combined with serious medical diseases
* Spinal cord injury, paraplegia
* The doctor or nurse believes that it is not appropriate to enroll patients (such as unable to cooperate in completing the study, unable to communicate effectively, severe mental anxiety, lower limb movement disorders, etc.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who come to our hospital and meet the inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
COST | Up to 12 months
  Perioperative cost
Visual Analogue Scale | Up to 12 months
  The basic method is to use a moving ruler with a length of about 10cm. One side is marked with 10 scales. The two ends are respectively "0" and "10" points. A point of 0 means no pain, and a point of 10 means the most intolerable Severe pain.
Oswestry Disability Index | Up to 12 months
  The minimum score for each item is 0 points, and the highest score is 5 points. The higher the score, the more severe the degree of dysfunction; the corresponding scores of the 10 items are accumulated. Calculate the percentage of the highest score (50 points) of the 10 items, which is the Oswestry dysfunction index. The higher the score, the more severe the patient's dysfunction.
modified Japanese orthopaedic association score | Up to 12 months
  Spinal function scoring method, including limb movement, sensory and bladder function evaluation, a total of 17 points. The higher the score, the better the recovery of spinal cord function.
SF-36(Medical Outcomes Study Short-Form 36) | Up to 12 months
  Medical Outcomes Study S hort-Form 36. There are 8 dimensions to evaluate health-related life quality (HRQOL), which are divided into two categories: physical health and physical health, namely physical function (PF), physical function (RP), physical pain (BP), General health (CH), vitality (VT), social function (SF), emotional function (RE), mental health (MH). The score is between 0-100, a high score indicates a good health.

SECONDARY OUTCOMES:
operation time | During surgery
  operation time
blood lose | During surgery
  blood lose
Radiation dose | During surgery
  Radiation dose
Complications | immediately after the surgery, up to 12 weeks
  Complications
Hospital stay | days between in and out hospital
  total hospital stay days
Deviation of screw | up to 12 months
  The deviation between the actual position of screw and the preoperative designed position

CONTACTS AND LOCATIONS:
Overall Officials: tian wei, MD,PHD, Study Chair — Beijing Jishuitan Hospital
Locations (1):
- Beijing Jishuitan hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
not decided